CLINICAL TRIAL: NCT00305877
Title: An Intergroup Randomized Phase II Study of Bevacizumab (NSC 704865) or Cetuximab (NSC 714692) in Combination With Gemcitabine and in Combination With Chemoradiation (Capecitabine and Radiation) in Patients With Completely-Resected Pancreatic Carcinoma
Brief Title: Bevacizumab or Cetuximab And Gemcitabine Hydrochloride, Capecitabine, and Radiation Therapy in Treating Patients With Pacreatic Cancer That Has Been Completely Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02969; NCI-2012-02969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-ECOG-E2204; SWOG-ECOG-E2204; ECOG-E2204; NCCTG-ECOG-E2204; E2204 (Other: Eastern Cooperative Oncology Group); E2204 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-12

CONDITIONS: Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine; Capecitabine; Radiotherapy; Radiation; Bevacizumab

ARMS (2):
- Arm I (cetuximab, gemcitabine, capecitabine, radiation) (Experimental): Patients receive cetuximab IV over 60-120 minutes on day 1, once weekly, in weeks 1-24; gemcitabine hydrochloride IV over 30 minutes on day 1, once weekly, in weeks 1-3, 13-15, 17-19, and 21-23; oral capecitabine twice daily on days 1-5, 5 days a week, in weeks 5-10. Patients also undergo radiotherapy once daily, 5 days a week, beginning in week 5 and continuing for approximately 5½ weeks (25 fractions).
  Interventions: Biological: cetuximab; Drug: gemcitabine hydrochloride; Drug: capecitabine; Radiation: radiation therapy; Other: laboratory biomarker analysis
- Arm II (bevacizumab, gemcitabine, capecitabine, radiation) (Experimental): Patients receive bevacizumab IV over 60-90 minutes on day 1 in weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23. Patients also receive gemcitabine hydrochloride and capecitabine and undergo radiotherapy as in arm I.
  Interventions: Drug: gemcitabine hydrochloride; Drug: capecitabine; Radiation: radiation therapy; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Arm I (cetuximab, gemcitabine, capecitabine, radiation)
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm II (bevacizumab, gemcitabine, capecitabine, radiation)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying bevacizumab to see how well it works compared to cetuximab when given together with gemcitabine, capecitabine, and radiation therapy in treating patients with pancreatic cancer that has been completely removed by surgery. Monoclonal antibodies, such as bevacizumab and cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bevacizumab or cetuximab together with gemcitabine, capecitabine, and radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether bevacizumab is more effective than cetuximab when given together with gemcitabine, capecitabine, and radiation therapy in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the toxicity profile of cetuximab and bevacizumab when combined with gemcitabine, before and after capecitabine plus radiation and during capecitabine plus radiation in patients with completely-resected pancreatic carcinoma in the adjuvant setting.

II. To assess the safety profile of either cetuximab or bevacizumab plus gemcitabine in patients with resected pancreatic cancer.

III. To obtain tissue specimens from resections of patients enrolled on study for correlative studies and further evaluations.

SECONDARY OBJECTIVES:

I. To evaluate disease-free and overall survival for patients receiving either cetuximab or bevacizumab in combination with gemcitabine before and after capecitabine plus radiation.

II. To assess the safety profile for patients receiving either capecitabine plus cetuximab plus radiation, or capecitabine plus bevacizumab plus radiation.

III. To correlate changes in serum amphiregulin and TGF alpha to survival, DFS and rash for patients receiving cetuximab.

IV. To determine the 2-year survival rate for patients receiving either cetuximab plus gemcitabine before and after capecitabine plus cetuximab plus radiation, or bevacizumab plus gemcitabine before and after capecitabine plus bevacizumab plus radiation.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to degree of prior resection of the pancreatic tumor (R0 vs R1). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive cetuximab IV over 60-120 minutes on day 1, once weekly, in weeks 1-24; gemcitabine hydrochloride IV over 30 minutes on day 1, once weekly, in weeks 1-3, 13-15, 17-19, and 21-23; oral capecitabine twice daily on days 1-5, 5 days a week, in weeks 5-10. Patients also undergo radiotherapy once daily, 5 days a week, beginning in week 5 and continuing for approximately 5½ weeks (25 fractions).

Arm II: Patients receive bevacizumab IV over 60-90 minutes on day 1 in weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23. Patients also receive gemcitabine hydrochloride and capecitabine and undergo radiotherapy as in arm I.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed evidence of pancreatic carcinoma
* Patients must have had all gross disease resected (R0 or R1 resection)
* Patients undergoing an R2 resection are not eligible
* Patients must have had no prior chemotherapy or radiation therapy for pancreatic cancer and must have had no prior EGFR/VEGF inhibition
* Patient must have ECOG performance status of 0-2
* Leukocytes >= 3,000/μL
* ANC >= 1,500/μL
* Platelets >= 100,000/μL
* Total bilirubin Within normal institutional limits
* AST (SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine clearance >= 60 mL/min for patients with creatinine levels above institutional normal
* Patients must be > 4 weeks and =< 8 weeks post-surgery at time of study registration (may be up to 10 weeks post-surgery prior to start of study therapy)
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception prior to study entry
* Women must not be pregnant or breast-feeding; all agents used in this study as well as radiation therapy to the abdomen have the potential for teratogenic or abortifacient effects; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Patients must not be receiving any other investigational agents
* Patients with known metastases are not eligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab, bevacizumab or other agents used in the study are not eligible
* Patients with wounds that have not fully healed are not eligible
* Patients must not have cardiac arrhythmia
* Patients must have no known HIV infection
* Patients must not have any of the following: acinar cell carcinoma, neuroendocrine carcinoma, cystadenocarcinoma, carcinosarcoma
* Patients with psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude them from meeting the study requirements are not eligible
* Patients requiring full dose anticoagulation are not eligible
* Patients with a history of transient ischemic attack (TIA) or cerebrovascular accident (CVA) are not eligible
* Patients with a history of the following within twelve months of study entry are not eligible:

  * Arterial thrombembolic events
  * Unstable angina
  * Myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on February 17, 2006 and terminated on January 9, 2008 with final accrual of 137 patients.
Groups:
- Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation): Patients receive cetuximab IV over 60-120 minutes on day 1, once weekly, in weeks 1-24; gemcitabine hydrochloride IV over 30 minutes on day 1, once weekly, in weeks 1-3, 13-15, 17-19, and 21-23; oral capecitabine twice daily on days 1-5, 5 days a week, in weeks 5-10. Patients also undergo radiotherapy once daily, 5 days a week, beginning in week 5 and continuing for approximately 5½ weeks (25 fractions).
- Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation): Patients receive bevacizumab IV over 60-90 minutes on day 1 every other week for 24 weeks. Patients also receive gemcitabine hydrochloride and capecitabine and undergo radiotherapy as in Arm A.
Period: Overall Study
Arm/Group | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation)
Started | 69 | 68
Treated | 67 | 63
Eligible | 66 | 66
Included in Efficacy Analysis | 65 | 62
Completed | 45 | 34
Not Completed | 24 | 34
Not completed — Lack of Efficacy | 6 | 9
Not completed — Adverse Event | 9 | 14
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Never start treatment | 2 | 5
Not completed — Ineligible | 2 | 1
Not completed — Transportation issue with daily RT | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation) | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Median (Full Range); unit: years] | 60 [29.2 to 92.9] | 60 [41.6 to 79.4] | 60 [29.2 to 92.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 65
  Male | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Specific Protocol Defined Adverse Event at Conclusion of All Therapy
Description: Specific toxicities to be monitored pursuant to the primary endpoint include:
  1. Any grade 5 toxicities
  2. Grade 4 dyspnea, neutropenic fever, allergic reaction, rash, wound dehiscence, wound infection, hypertension
  3. Grade 3 or higher arterial thromboembolic phenomena, bleeding, phlebitis/deep vein thrombosis (DVT)/pulmonary embolism (PE), hemorrhage, ileus, bowel perforation, diarrhea, and mucositis
  4. ECOG performance status decline by 2 or greater for >24 hours
  5. Weight loss >10%
Time Frame: Every 2 weeks while on treatment and for 30 days after the end of treatment
Population: All treated patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation)
Number analyzed (Participants) | 67 | 63
Proportion of patients | 0.30 [0.19 to 0.42] | 0.25 [0.15 to 0.38]

2. Secondary Outcome: Two-year Overall Survival Rate
Description: Overall survival (OS) is defined as the time from randomization to death from any cause, or censored at last known date of survival.
Time Frame: Assessed every 3 months for 2 years
Population: Eligible and treated patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation)
Number analyzed (Participants) | 65 | 62
Proportion of patients | 0.38 [0.26 to 0.50] | 0.37 [0.24 to 0.48]

3. Secondary Outcome: Two-year Disease-free Survival (DFS)
Description: Disease-free survival (DFS) is defined as the time from randomization to the first treatment failure (recurrence or death before recurrence).
Time Frame: Assessed every 3 months for 2 years, and every 6 months after completion of treatment for 2 years, then annually for 3 years
Population: Eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation)
Number analyzed (Participants) | 65 | 62
Proportion of patients | 0.17 [0.08 to 0.26] | 0.23 [0.12 to 0.34]

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation)
Serious Adverse Events (participants affected / at risk) | 54/67 | 51/63
Other Adverse Events (participants affected / at risk) | 66/67 | 60/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) (N=67) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation) (N=63)
Allergic reaction (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 4
Leukocytes decreased (Investigations) | 25 | 24
Lymphopenia (Investigations) | 10 | 7
Neutrophils decreased (Investigations) | 29 | 35
Platelets decreased (Investigations) | 4 | 9
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
C-P arrest, non-fatal, cause unknown (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Fatigue (General disorders) | 11 | 6
Rigors/chills (General disorders) | 0 | 1
Weight loss (Investigations) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 4
Ascites (non-malignant) (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Perforation, colon (Gastrointestinal disorders) | 0 | 1
Ulcer, gastric (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Hepatic-other (Hepatobiliary disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, biliary tree (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, catheter (Infections and infestations) | 2 | 0
Infection Gr0-2 neut, peritoneal (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 | 0
Infection w/ unk ANC liver (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, blood (Infections and infestations) | 1 | 0
Infection-other (Infections and infestations) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2
Alkaline phosphatase increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Creatinine increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Abdomen, pain (Gastrointestinal disorders) | 0 | 4
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cetuximab, Gemcitabine, Capecitabine, Radiation) (N=67) | Arm B (Bevacizumab, Gemcitabine, Capecitabine, Radiation) (N=63)
Anemia (Blood and lymphatic system disorders) | 28 | 28
Leukocytes decreased (Investigations) | 47 | 39
Lymphopenia (Investigations) | 12 | 4
Neutrophils decreased (Investigations) | 34 | 34
Platelets decreased (Investigations) | 36 | 34
Hypertension (Vascular disorders) | 1 | 16
Hypotension (Vascular disorders) | 4 | 1
Fatigue (General disorders) | 49 | 48
Fever w/o neutropenia (General disorders) | 16 | 10
Insomnia (Psychiatric disorders) | 6 | 0
Rigors/chills (General disorders) | 8 | 7
Weight loss (Investigations) | 17 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 12
Nail changes (Skin and subcutaneous tissue disorders) | 11 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 21 | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 56 | 10
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 27 | 9
Skin-other (Skin and subcutaneous tissue disorders) | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 30 | 19
Constipation (Gastrointestinal disorders) | 14 | 11
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 34 | 29
Dyspepsia (Gastrointestinal disorders) | 5 | 8
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 21 | 9
Nausea (Gastrointestinal disorders) | 43 | 38
Taste disturbance (Nervous system disorders) | 11 | 5
Vomiting (Gastrointestinal disorders) | 28 | 13
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Edema limb (General disorders) | 7 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 32 | 18
Alkaline phosphatase increased (Investigations) | 27 | 15
Alanine aminotransferase increased (Investigations) | 26 | 20
Aspartate aminotransferase increased (Investigations) | 32 | 24
Blood bilirubin increased (Investigations) | 5 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 19 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 18 | 0
Hypokalemia (Metabolism and nutrition disorders) | 13 | 5
Proteinuria (Renal and urinary disorders) | 1 | 8
Hyponatremia (Metabolism and nutrition disorders) | 9 | 3
Dizziness (Nervous system disorders) | 9 | 2
Neuropathy-motor (Nervous system disorders) | 5 | 0
Neuropathy-sensory (Nervous system disorders) | 5 | 4
Abdomen, pain (Gastrointestinal disorders) | 22 | 21
Head/headache (Nervous system disorders) | 7 | 9
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Flu-like syndrome (General disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less